CLINICAL TRIAL: NCT05897424
Title: A Phase 2, Single Arm, Open Label Extension Study, Evaluating the Long-Term Safety and Clinical Efficacy of SAR447537 (INBRX-101) in Adults With Alpha-1 Antitrypsin Deficiency (AATD) Emphysema
Brief Title: Long-term, Open-label Study of SAR447537 (INBRX-101) in Adults With Alpha-1 Antitrypsin Deficiency Emphysema
Acronym: ELEVAATE OLE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INBRX101-01-202; 2023-508137-14-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Alpha 1-Antitrypsin Deficiency; Emphysema
Keywords: AATD; Alpha 1-Antitrypsin Deficiency; Emphysema; INBRX-101; AAT; SAR447537
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema

STUDY DESIGN:
Intervention Model Description: Multicenter, single arm, open-label extension study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SAR447537 (INBRX-101) (Experimental): A1PI, Recombinant, Bivalent Fc Fusion Protein, in a solution for intravenous injection
  Interventions: Drug: SAR447537

INTERVENTIONS:
Drug: SAR447537 — A1PI, Recombinant, Bivalent Fc Fusion Protein

SUMMARY:
Phase 2 open label extension study to evaluate SAR447537 (INBRX-101) in adults with AATD emphysema

DETAILED DESCRIPTION:
This is a Phase 2, Single Arm, Open Label Extension Study, Evaluating the Long-Term Safety and Clinical Efficacy of SAR447537 (INBRX-101) in Adults With Alpha-1 Antitrypsin Deficiency (AATD) Emphysema.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18-80 years of age, inclusive, at the time of screening
2. Diagnosis of AATD
3. Evidence of emphysema secondary to AATD
4. FEV1 of ≥ 30% predicted at screening and post-bronchodilator FEV1/FVC<0.7
5. Current non-smoking status

Exclusion Criteria:

For newly identified participants

1. Receipt of A1PI augmentation therapy within 5 weeks prior to the first dose of study drug
2. Known or suspected allergy to components of SAR447537, A1PI or human IgG
3. Uncontrolled diabetes mellitus despite adequate antidiabetic pharmacologic treatment with a screening HbA1c value ≥9%
4. Received IV immunoglobulins, monoclonal antibodies and/or other biologic therapies within 30 days
5. On waiting list for lung or liver transplant
6. Acute respiratory tract infection or COPD exacerbation within 4 weeks prior to or during screening
7. Evidence of decompensated cirrhosis
8. Active cancers or has a history of malignancy within 5 years prior to screening
9. History of unstable cor pulmonale

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Long-term safety and tolerability | 3 years
  Incidence of all treatment emergent adverse events (TEAEs), TEAEs ≥ Grade 3, serious adverse events (SAEs), TEAEs leading to discontinuation from SAR447537, and adverse events of special interest (AESIs) (including infusion-related reactions).

SECONDARY OUTCOMES:
Change in lung density by quantitative computerized tomography (CT) | 3 years
  Assess the annual rate of change in lung density assessed by serial quantitative CT (15th percentile point, PD15) at total lung capacity (TLC), centrally read, from baseline to end of treatment (EoT).
Trough SAR447537 concentration changes | 3 years
  Change in SAR447537 concentration levels from baseline to end of treatment
Trough serum functional AAT (fAAT) concentration changes | 3 years
  Change in fAAT concentration levels from baseline to end of treatment
Covariate Analysis: Biometric Values: Weight | 3 years
  Assessment of the impact of participant's weight [in kg] on the pharmacokinetic profile of SAR447537
Covariate Analysis: Biometric Values: Height | 3 years
  Assessment of the impact of participant's height [in cm] on the pharmacokinetic profile of SAR447537
Covariate Analysis: Biometric Values: Age | 3 years
  Assessment of the impact of participant's age [in years] on the pharmacokinetic profile of SAR447537
Covariate Analysis: Biometric Values: Sex | 3 years
  Assessment of the impact of participant's sex [male or female] on the pharmacokinetic profile of SAR447537
Anti-drug antibodies | 3 years
  Frequency of anti-drug antibodies (ADA) against SAR447537 as well as neutralizing ADA (NAb) against SAR447537

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (40):
- United States (18):
  - UAB Lung Health Center- Site Number : 105, Birmingham, Alabama
  - St Joseph's Hospital and Medical Center- Site Number : 126, Phoenix, Arizona
  - David Geffen School of Medicine at UCLA- Site Number : 124, Los Angeles, California
  - University of California Davis Medical Center- Site Number : 110, Sacramento, California
  - National Jewish Medical and Research Center- Site Number : 123, Denver, Colorado
  - Nuvance Health Medical Practices, Pulmonary & Sleep Specialists- Site Number : 119, Danbury, Connecticut
  - University of Florida - Gainesville - 1600 SW Archer Rd- Site Number : 101, Gainesville, Florida
  - Indiana University- Site Number : 127, Indianapolis, Indiana
  - Brigham and Women's Hospital -75 Francis Street- Site Number : 131, Boston, Massachusetts
  - University of Minnesota-420 Delaware Str SE- Site Number : 125, Minneapolis, Minnesota
  - Hannibal Regional Healthcare System-HRMG-Hannibal- Site Number : 111, Hannibal, Missouri
  - Columbia University Irving Medical Center- Site Number : 104, New York, New York
  - Oregon Health and Science University- Site Number : 117, Portland, Oregon
  - Penn State Health Milton S. Hershey Medical Center- Site Number : 122, Hershey, Pennsylvania
  - Temple University Hospital - 3401 N Broad St- Site Number : 130, Philadelphia, Pennsylvania
  - Velocity Clinical Research - Spartanburg - PPDS- Site Number : 120, Spartanburg, South Carolina
  - Houston Methodist Hospital- Site Number : 113, Houston, Texas
  - University of Utah Health Care- Site Number : 106, Salt Lake City, Utah
- Australia (6):
  - Investigational Site Number : 202, Chermside, Queensland
  - Investigational Site Number : 204, South Brisbane, Queensland
  - Investigational Site Number : 201, North Adelaide, South Australia
  - Investigational Site Number : 207, Box Hill, Victoria
  - Investigational Site Number : 203, Fitzroy, Victoria
  - Investigational Site Number : 205, Frankston, Victoria
- Denmark (2):
  - Investigational Site Number : 701, Hellerup
  - Investigational Site Number : 702, Vejle
- Investigational Site Number : 501, Dublin, Dublin, Ireland
- New Zealand (2):
  - Investigational Site Number : 403, Auckland
  - Investigational Site Number : 404, Wellington
- Poland (2):
  - Investigational Site Number : 801, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 802, Krakow
- Spain (3):
  - Investigational Site Number : 901, Santander, Cantabria
  - Investigational Site Number : 902, Madrid
  - Investigational Site Number : 903, Santiago de Compostela
- Investigational Site Number : 601, Gothenburg, Sweden
- United Kingdom (5):
  - Investigational Site Number : 308, Dundee, Angus
  - Investigational Site Number : 306, Wythenshawe, Cheshire
  - Investigational Site Number : 307, Exeter, Devon
  - Investigational Site Number : 304, Southampton, Hampshire
  - Investigational Site Number : 309, Coventry

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: INBRX101-01-202 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26402&tenant=MT_SNY_9011